CLINICAL TRIAL: NCT06486597
Title: Whole Body Metabolism in Children With Cerebral Palsy With Low Skeletal Muscle Mass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Cathrine Oerngreen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-B01-1066
Record Dates: First submitted 2024-05-17; First posted 2024-07-03 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Meal intervention with stable isotopes (Experimental): A liquid mixed meal are gived adjusted by weight. The meal consists of: Intrinsically labelled D5-Phenylalanine and D3-Leucine labelled casein protein, 13C16palmitate, 13C6-Glucose in a mix of glucose, casein protein and rape seed oil dissolved in water in an energy density of 50% CHO, 35% fat and 15% protein. Blood samples are drawn frequently to measure fat, glucose and protein metabolism.
  Interventions: Dietary Supplement: Meal

INTERVENTIONS:
Dietary Supplement: Meal — Liquid meal

SUMMARY:
At the center of pediatrics in Copenhagen the investigators experience that the children with CP with low skeletal muscle mass have more complications and admission after for example surgery is prolonged due to these complications. In order to prevent malnutrition and energy insufficiency as well as obesity and cardiometabolic disorders in adulthood, and with the aim of defining biomarkers for energy needs, the investigators wish to determine energy and protein needs in children with CP.

The investigators wish to investigate the whole-body metabolism in children with cerebral palsy (CP) and compare the results with results from healthy children. The investigators aim to include 10 children (aged 2-18 years) with CP with low skeletal muscle mass and 10 healthy controls (aged 2-18 years). By using stable isotope technique the investigators will investigate systemic fat, glucose and protein metabolism together with liver protein degradation and glucose production. Furthermore, by using DXA scan the investigators will describe the quality and distribution of skeletal muscle. Lastly, the investigators will determine the skeletal muscle signal pathway and metabolism in skeletal muscle via the Bergström biopsy technique in vastus lateralis.

DETAILED DESCRIPTION:
Trial design and time frame:

A prospective, non-randomized, cross-sectional study.

There will be two different groups included:

* Children with cerebral palsy with low skeletal muscle mass
* Healthy controls: Children admitted to the hospital at the Epilepsy monitor unit (EMU for conditions not affecting metabolic function)

The trial will be conducted over a total of five days and takes place at the Copenhagen Neuromuscular Centre, Department of Neurology or Department of Pediatrics and Adolescent Medicine, Rigshospitalet

Study Day 1: The patient will be DXA-scanned or fat mass will be measured by a fat caliper, and the patient will complete quality of life questionnaire and pain scores.

Study Day 2 (Study type A): The stable isotope infusion will take place. The subjects will arrive around 08.00, at Copenhagen Neuromuscular Centre (CNMC), Rigshospitalet or Department of Pediatrics and Adolescents medicine, Rigshospitalet. Otherwise, the study will take place when the child is admitted for change of baclofen pump or minor surgery, where they typically will be hospitalized for 1-3 days at Rigshospitalet or Skejby hospital at the Department of Pediatrics and Adolescents or the Orthopedic Departments.

On arrival, EMLA (local anesthetics cream) will be applied on the skin of the children to minimize any discomfort that may occur during IV-insertion. Two peripheral venous catheters are inserted, one in the medial cubital vein for infusion of stable isotopes, and one in a dorsal vein of the hand for blood sampling. Most of the children already have a permanent catheter, and in this case the permanent catheter will be used for infusion of stable isotopes.

Background samples will be collected before the start of tracer infusion. After 1 hour and 45 minutes of basal tracer infusion, basal blood samples are drawn (time -15 and -30) for the determination of basal steady state tracer enrichments and hormone concentrations. At time= 0, a liquid mixed meal is provided. Blood samples are drawn regularly for 6 hours and more frequently the first hour after the test meal ingestion (at 0, 10, 20, 30, 40, 50, 60, 90, 120, 180, 240, 300 and 360 minutes). If the child becomes upset or the investigators for other reasons want to stop earlier than 6 hours, the already obtained blood and urine samples will be analyzed and included in the results.

Study days 3, 4, and 5 (Study type B and C):

These study days are optional to the families and the investigator. For some families one study day is what they can fit into their calendar, and the investigators want to respect that, for those who accept to continue the study for more than one day, the following days are included.

The doubly labeled water technique measures energy consumption over a prolonged period, in our study for 1 week. A drink with doubly labeled water will be ingested, and energy expenditure is measured by urine and blood sampling. This method is repeated at 3 hours and 4 hours after the drink intake and again at day 3 and day 7. Furthermore, a drink with 13C will be ingested, and breath tests collected in vacutainers with straws will be collected for analysis of energy expenditure. Measuring energy expenditure with these two less non-invasive methods and comparing results with the detailed meal test, will pave the way for developing simple diagnostic markers for metabolism in the children.

The tracers: In this study, the investigators will intravenously infuse small amounts of metabolites labelled with stable isotopes in primed continuous intravenous infusions of: D8-Phenylalanine, D2-Tyrosine, 13C18-Oleate acid, D2-Glucose, D5-Glycerol. This method is well-established at both CIMT and CNMC and has been used investigating several of patients categories before: Neonates (ongoing study), gastric sleeve, elderly and neuromuscular patients.

The tracers are prepared from the hospital pharmacy. All tracers are purchased from Cambridge Isotope Laboratories, Andover, MA, USA suitable for human use. Stable isotopes are non-radioactive and naturally occurring in food (e.g. in corn).

Food intervention: At time= 0 (120 minutes after infusion), a liquid mixed meal adjusted by weight is given. The meal consists of: Intrinsically labelled D5-Phenylalanine and D3-Leucine labelled casein protein, 13C16palmitate, 13C6-Glucose in a mix of glucose, casein protein and rape seed oil dissolved in water in an energy density of 50% CHO, 35% fat and 15% protein. Intrinsically labeled caseinate was produced via an infusion of [D5]-phenylalanine and [D3]leucine into a lactating cow to obtain enriched milk Foulumn, Arhus University, from which the caseinate fraction was isolated at Arla Foods according to Good Manufacturing Practice (GMP) and safety checked an store under appropriate regulatory conditions until use (Nørre Vium, Denmark) following a previously described procedure.

Analyses of blood samples:The samples will be collected in syringes containing 10μL EDTA/mL to prevent coagulation. The blood is immediately centrifuged at 4oC to separate plasma from red blood cells. The samples will be frozen in coded tubes and stored at -80C until analysis.

Routine blood samples: Will be analysed immediately at the Department of Clinical Biochemistry, Rigshospitalet:

- Blood samples include: Insulin, HbA1C, Cholesterol, HDL, LDL, triglycerides

Glucose and lactate: will be analyzed (ABL 700) immediately as the blood is drawn.

Specific blood samples:

Free fatty acids: will be analyzed using fluorometry. Hormones (catecholamines, insulin, incretins and glucagon): will be analyzed using RIA and Elisa Methods respectively. Stable isotope enrichments in blood: will be analyzed using Liquid chromatography-tandem mass-spectrometry (LC-MS/MS) and gas chromatography combustion isotope ratio mass spectrometry (GC-C-IRMS) (Thermo Scientific, Palo Alto, CA, USA and Bremen, Germany). Calculations: Whole body metabolite quantitative kinetics will be calculated using Steele's equation for non-steady state adapted for analysis of stable isotopes under the post-absorptive conditions.

ELIGIBILITY:
Inclusion Criteria:

* -Children with cerebral palsy with low skeletal muscle mass

  o Being wheelchair dependent GMFCS IV-V
* Healthy controls: Children admitted to the EMU because of either

  * Classification of epilepsy or to rule out differential diagnoses of epilepsy
  * Nocturnal EEG changes

Age:

o 2-18 years

- Signed informed consent to participation in the trial.

Exclusion Criteria:

* Inability to understand the purpose of the trial or cooperate in the conduction of the experiments. For the children this will concern of course the parents or the guardians of the child.
* Competing conditions at risk of compromising the results of the study.
* In healthy children, concerns that participation in the trial may affect the diagnostic quality of the EMU investigation
* Participation in other trials that may interfere with the results.
* Intake of medications that may interfere with the results, evaluated by investigator.
* Pregnancy or breastfeeding.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Protein breakdown | 10 hours
  Phenylalanine Rate of appearance micro mol/kgFFM/min in a fasted and fed state

SECONDARY OUTCOMES:
Muscle biopsy | 10 hours
  Muscle morphology
Life quality score | 10 hpurs
  Life quality score by using Pediatric Quality of Life Inventory (PedsQL) (0-100), high score indicates worse qualiity of life.
Quality of Skeletal Muscle | 10 hours
  Dual-energy X-ray absorptiometry (DEXA) scan
Metabolities | 10 hours
  Concentration of plasma amino acids (mmol/L), concentration of glucose (mmol/L), concentration of palmitate (micromol/L), concentration of free fatty acids (mmol/L) and levels of HbA1c (mmol/mol)
Hormones | 10 hours
  Concentration of Insulin (pmol/L), concentration of catecholamines (nmol/l) , glucagon (pmol/L), gut hormones and incretins (GLP-1 (pmol/L) and GIP, (pmol/L))
Energy utilization | 10 hours
  Energy expenditure assessed by doubly labeled water method and 13C breath test to test that these methods are valuable and can be used in the future as less expensive and invasive methods to measure energy utilization.
Muscle biopsy | 10 hours
  muscle fiber type
muscle biopsy | 10 hours
  size
Muscle biopsy | 10 hours
  Protein markers: MuRF1, MAFbx, FoxO (ng/mg total protein)
Muscle biopsy | 10 hours
  muscle generating markers: Myo D, Myogenin, IGF1 (ng/mg total protein )
Muscle biopsy | 10 hours
  Muscle growth regulating protein (myostatin)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics and Adolescent Medicine and Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark